CLINICAL TRIAL: NCT06684093
Title: Effects of Back Squat Exercise with or Without Blood Flow Restriction in Healthy Adolescent Basketball Athletes: a Randomized Controlled Trial
Brief Title: Effects of Back Squat Exercise with or Without Blood Flow Restriction in Healthy Adolescent Basketball Athletes
Acronym: BFR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St Joseph University, Beirut, Lebanon (Other)
Responsible Party: Principal Investigator, Perla Mjaess, Study coordinator, St Joseph University, Beirut, Lebanon
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2023-325
Record Dates: First submitted 2024-10-17; First posted 2024-11-12 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Adolescent Athletic Performance; Muscle Strength Development; Jump Height Improvement; Ground Reaction Force (GRF) Enhancement; Injury Prevention in Sports; Blood Flow Restriction (BFR) Training Effects; Reduced Mechanical Load on Joints
Keywords: Blood Flow Restriction training; high intensity training; basketball; injury prevention; jump height; ground reaction force

STUDY DESIGN:
Intervention Model Description: The study uses a Parallel Assignment model where participants are randomly assigned to one of two intervention groups.
  Group 1: Blood Flow Restriction (BFR) Training Group - Participants engage in low-load resistance training (20-30% of 1-repetition maximum) with blood flow restriction applied to the working muscles using pressure cuffs. The training focuses on strengthening the quadriceps, hamstrings, and calf muscles.
  Group 2: Traditional High-Intensity Training Group - Participants perform high-intensity resistance exercises (70-85% of 1-repetition maximum) targeting the same muscle groups as the BFR group.
  Both groups undergo the respective training protocols three times a week over 8-12 weeks. Performance outcomes, including muscle strength, jump height, and ground reaction force (GRF), are measured at baseline, mid-intervention, and post-intervention. The parallel assignment allows a direct comparison of the effects of BFR training versus traditional high-intensity training on
Who Masked: Outcomes Assessor
Masking Description: In this study, only the Outcomes Assessor is masked to the group assignments. The assessors responsible for measuring muscle strength, jump height, and ground reaction force (GRF) are unaware of which participants belong to the Blood Flow Restriction (BFR) training group or the traditional high-intensity training group. This masking aims to minimize bias during the evaluation and analysis of performance outcomes. The participants, care providers, and investigators are aware of the group assignments, as they are directly involved in the delivery and participation in the specific training protocols.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Back Squat Exercise without Blood Flow Restriction (Active Comparator): In this arm of the study, participants will perform back squat exercises without any blood flow restriction. This group serves as a control to evaluate the effects of traditional resistance training alone on strength and muscle development in healthy adolescent basketball athletes.
  Interventions: Behavioral: Back squats
- Back Squat Exercise with Blood Flow Restriction (Experimental): This arm of the study involves participants performing back squat exercises while blood flow restriction is applied to the upper legs. The aim is to assess the effects of combining traditional resistance training with blood flow restriction on strength and muscle hypertrophy in healthy adolescent basketball athletes.
  Interventions: Device: Back squat with Blood flow restriction machine

INTERVENTIONS:
Device: Back squat with Blood flow restriction machine — The blood flow restriction (BFR) machine is a specialized device designed to safely apply controlled pressure to the proximal limbs during exercise. It typically consists of adjustable cuffs or bands that are placed around the upper arms or thighs, which are connected to a pressure monitoring system. The device enables practitioners to restrict venous blood flow while allowing arterial blood flow to the working muscles. This method enhances the effects of low-intensity resistance training by promoting muscle hypertrophy and strength gains, similar to those achieved through high-intensity training. The BFR machine is commonly used in rehabilitation settings and athletic training programs to optimize performance and recovery while minimizing the risk of injury.
  Arms: Back Squat Exercise with Blood Flow Restriction
Behavioral: Back squats — Back squats without any blood flow restriction
  Arms: Back Squat Exercise without Blood Flow Restriction

SUMMARY:
The goal of this clinical trial is to assess the effectiveness of Blood Flow Restriction (BFR) training compared to traditional high-intensity training in adolescent basketball players aged 16-18. The main questions it aims to answer are:

Does BFR training improve muscle strength more effectively than traditional high-intensity training? Does BFR training enhance jump height and ground reaction force (GRF) while reducing mechanical load? Researchers will compare BFR training to traditional high-intensity training to see if BFR training offers greater improvements in muscle strength, jump height, and GRF while potentially reducing knee joint stress.

Participants will:

Be randomly assigned to either the BFR training group or the high-intensity training group.

Undergo performance evaluations, including measurements of muscle strength, jump height, and GRF at three time points throughout the study.

Follow a training protocol specific to their assigned group

DETAILED DESCRIPTION:
Detailed Description:

This randomized controlled study aims to evaluate the effectiveness of Blood Flow Restriction (BFR) training compared to traditional high-intensity training in adolescent basketball players, focusing on performance enhancement and safety. The study was approved by the Committee Research Ethics of Saint Joseph University of Beirut (Code: 2023-325) on December 7, 2023.

Study Setting and Participants: The research was conducted within two sports academies in Lebanon, Mont La Salle and Rebound academies. A total of 50 adolescent basketball players, aged 16-18 years, participated. Inclusion criteria required regular training (at least three sessions per week) and competitive basketball experience within the last six months. Exclusion criteria included history or presence of cardiovascular, pulmonary, or metabolic conditions, vascular disorders, coagulation disorders, or ongoing anticoagulant therapy. Before starting the study, participants completed a recruitment questionnaire to gather demographic data and assess eligibility for BFR training.

Study Design and Randomization: Participants were randomly assigned into two groups:

Group 1 (BFR Training Group): Engaged in low-intensity resistance training (20-30% of 1RM) with BFR using pressure cuffs on the lower limbs.

Group 2 (High-Intensity Training Group): Engaged in traditional high-intensity resistance training (65-80% of 1RM) without BFR.

Both groups completed 12 sessions over six weeks, with a 48-hour interval between sessions. The study's structured approach allows for a comparison of the training modalities' effects on muscle strength, jump height, and ground reaction force (GRF).

Evaluation Protocol: Participants underwent baseline assessments before starting the exercise regimen. These assessments included occlusion pressure, 1-repetition maximum (1RM) testing, muscle strength, jump height, and GRF.

Occlusion Pressure Measurement: Measured using the VALD-performance system (Version 3 of the Airbands model, Australia) with athletes seated and cuffs placed proximally on the thigh (25% of the femur length).

1RM Testing: Participants performed warm-up sets before progressively increasing load until reaching the maximum weight they could lift with proper form.

Muscle Strength: Assessed using a digital dynamometer (KINVENT, K-PULL, France) for both quadriceps and hamstring muscles.

Jump Height and GRF: Evaluated using a force platform (KINVENT, France) during counter-movement jumps (CMJs).

Evaluations were conducted at three time points: baseline (M1), mid-intervention at three weeks (M2), and post-intervention at six weeks (M3). Each measurement was performed three times to ensure inter-rater reliability, with four physiotherapists maintaining consistency by evaluating the same athletes throughout the study.

Intervention Protocols:

Group 1 (BFR Training Group): Performed four sets of back squats at 20% of 1RM during weeks 1-3, increasing to 25% at week 3, and 30% during weeks 5-6.

Group 2 (High-Intensity Training Group): Began with 65% of 1RM in weeks 1-3, increasing to 70% at week 3, and 80% during weeks 5-6.

Both protocols aimed to progressively enhance strength while monitoring the effects on joint stress and overall performance.

Outcome Measures: The primary outcomes included changes in quadriceps and hamstring strength, jump height, and GRF over the intervention period. Secondary outcomes assessed knee joint stress and participant satisfaction with their respective training protocols.

Statistical Analysis: Data were analyzed using XLStat® software (AddinsoftR, Paris, France; version 2019.1.2). Descriptive statistics were calculated for demographic data. Mann-Whitney U tests were used for comparing groups, while Wilcoxon signed-rank tests evaluated within-group differences across time points (ΔM2-M1, ΔM3-M2, and ΔM3-M1). The reliability of measurements was assessed using the Intraclass Correlation Coefficient (ICC).

The study results are expected to provide insights into the effectiveness of BFR as a safer, low-load alternative to traditional high-intensity training in adolescent athletes, potentially offering a means to optimize performance while minimizing injury risk.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 16 and 18 years.
* Engaged in basketball training sessions at least three times per week.
* Competed in basketball within the last six months.
* No major injuries that limit their training session routines.

Exclusion Criteria:

* History or presence of cardiac, pulmonary, or metabolic conditions.
* Presence of vascular disorders in the upper or lower limbs.
* Individuals with coagulation disorders or those undergoing anticoagulant therapy.
* Recent surgeries or chronic conditions contraindicating Blood Flow Restriction (BFR) training.

Ages: 16 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 39 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
Quadriceps Muscle strength (Kg) | Baseline (Day 0, before starting the protocol), 3 weeks after baseline (Day 21), and 48 hours after the last session, approximately 6 weeks after baseline (Day 42).
  Assessed using a digital dynamometer, this measure reflects the improvement in quadriceps strength, a key indicator of the effectiveness of low-intensity training with BFR.

SECONDARY OUTCOMES:
Hamstring Muscle Strength (kg) | Baseline (Day 0, before starting the protocol), 3 weeks after the baseline assessment (Day 21), and 48 hours after the last session, approximately 6 weeks after the baseline assessment (Day 42).
  Evaluates the hamstring strength using a digital dynamometer to provide a broader view of muscle strength changes.
Jump Height (cm) | Baseline (Day 0), 3 weeks after baseline (Day 21), and 48 hours after the last session, approximately 6 weeks after baseline (Day 42).
  Measures maximum jump height using a force platform to assess changes in lower limb explosive power.
Ground reaction force (Newton) | Baseline (Day 0), 3 weeks after baseline (Day 21), and 48 hours after the last session, approximately 6 weeks after baseline (Day 42).
  Assesses the peak force generated during the landing phase of a countermovement jump using a force platform.

OTHER OUTCOMES:
1RM (One Repetition Maximum) (kg) | Baseline (Day 0), 3 weeks after baseline (Day 21), and 48 hours after the last session, approximately 6 weeks after baseline (Day 42).
  Evaluates the maximum weight that an athlete can lift in a single squat repetition.
Occlusion Pressure (mmHg) | Pre-exercise on Day 0 (Baseline).
  Measures the pressure applied during the BFR sessions, recorded using an automated system.
Inter-Rater Reliability (ICC) | Throughout the duration of the study (up to 6 weeks).
  Evaluates the reliability of the measurements performed by different physiotherapists using the Intraclass Correlation Coefficient (ICC).

CONTACTS AND LOCATIONS:
Locations (1):
- Two sports academies in Lebanon (Mont la salle and Rebound academies), Beirut, Lebanon

IPD SHARING:
Plan to Share IPD: Yes
In this study, the investigators plan to share the following specific individual participant data (IPD) upon completion of the trial:
  Demographic Information:
  Participants' age, gender, and baseline characteristics such as height, weight, and basketball experience.
  Intervention Details:
  Information regarding which intervention each participant received, specifically whether they performed back squat exercises with blood flow restriction or standard back squat exercises without restriction.
  Outcome Measures:
  Results for primary and secondary outcome measures, including:
  Muscle strength (1-repetition maximum testing results). Muscle hypertrophy (cross-sectional area measurements via ultrasound). Jump height Ground reaction force
  Adverse Events:
  Any recorded adverse events or side effects related to the interventions during the study period.
  Study Protocol Data:
  A summary of the study protocol, including the randomization process, assessment methods, and data collection procedures.
Supporting Information: Study Protocol, SAP, ICF